CLINICAL TRIAL: NCT03332485
Title: A Randomized, Investigator- and Colonoscopist-blinded, Phase 2 Study of the Efficacy and Safety of ECP (Polyethylene Glycol 3350 [PEG 3350]) Colon Prep Kit Compared With MoviPrep® Split-dose for Colonoscopy Preparation
Brief Title: Safety and Efficacy Study of an Edible Colonoscopy Preparation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sebela Pharmaceuticals Development LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SEB-ECP-202
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Colon Prep for Colonoscopy
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ECP Colon Prep Kit (Experimental)
  Interventions: Drug: ECP Colon Prep Kit
- MoviPrep® (Active Comparator)
  Interventions: Drug: MoviPrep®

INTERVENTIONS:
Drug: ECP Colon Prep Kit — ECP Colon Prep Kit
  Arms: ECP Colon Prep Kit
Drug: MoviPrep® — MoviPrep®
  Arms: MoviPrep®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ECP (PEG 3350) Colon Prep Kit compared with MoviPrep split-dose as a colon-cleansing preparation for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a medically indicated colonoscopy for colorectal cancer screening or surveillance for colorectal cancer
* Females must be non-lactating and have a negative pregnancy test if of child bearing potential
* Ability and willingness of subject to participate fully in all aspects of this clinical trial
* Written informed consent

Exclusion Criteria:

* Known or suspected clinically significant intestinal stricture of any etiology
* History of diabetes mellitus, controlled with insulin
* Taking insulin by injection
* Pregnant or lactating
* Renal insufficiency, hypokalemia, hyperkalemia, chronic liver disease or arrhythmic disorder
* Chronic heart failure or recent (within 90 days of screening) acute heart failure
* Receiving warfarin, heparin, clopidogrel, Pradaxa®, Xarelto®, Effient® or other blood thinning agents
* Short bowel syndrome
* Known diagnosis of Crohn's disease or ulcerative colitis, exclusionary only if subject has a history of any bowel resection, has suspected active inflammation, has symptoms suggestive of obstruction or a known bowel stricture
* Severe psychological disease causing functional impairment limiting capacity to complete the preparation
* Impaired consciousness increasing the risk of aspiration
* Used narcotics/opiates within the 14 days prior to the colonoscopy
* Used an anti-diarrheal within the 14 days prior to the colonoscopy procedure
* Uses drugs of abuse including abused prescription medication
* Used iron supplements within 14 days of the colonoscopy procedure
* History of gastrointestinal surgery other than appendectomy or cholecystectomy
* Diagnosis of gastroparesis or ileus
* Symptoms of chronic constipation defined as fewer than 3 bowel movements per week on average over the previous 3 months
* History of a failed bowel preparation, defined as either requiring an enema the day of the colonoscopy or needing to have the colonoscopy repeated
* CTCAE grade 1 sodium, potassium or magnesium at screening
* Clinically significant abnormalities (ketones, protein, glucose) at screening urinalysis, in the opinion of the investigator
* Any known allergies to any of the ingredients or ECP Colon Prep Kit (including coconut) or the active comparator
* Unable or unwilling to consume all components of the study drug including aversions to or adverse events from flavoring
* Received any investigational therapy within 30 days of initiation of study drug
* Serious underlying disease that, in the opinion of the investigator, may interfere with the subject's ability to participate fully in the study
* Requirement to use chromoendoscopy during the procedure for the purpose of surveillance for colorectal dysplasia or cancer in subjects with inflammatory bowel disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with successful bowel cleansing defined as centrally read 4 point modified Aronchick Scale (1=Inadequate, 2=Fair, 3=Good, 4=Excellent) score of either good or excellent. | 24-hour period, beginning the day prior to the procedure and through the morning of the colonoscopy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Hall, Study Director — Sebela Pharmaceuticals Development LLC
Locations (8):
- United States (8):
  - Sebela Site 007, Anaheim, California
  - Sebela Site 006, Indianapolis, Indiana
  - Sebela Site 002, Bastrop, Louisiana
  - Sebela Site 003, Annapolis, Maryland
  - Sebela Site 004, Great Neck, New York
  - Sebela Site 008, Wilmington, North Carolina
  - Sebela Site 001, Mentor, Ohio
  - Sebela Site 005, Ogden, Utah